CLINICAL TRIAL: NCT00169325
Title: Clinical, Neurophysiological and Radiological Evaluation of Patients With Basal Ganglia Lesions
Status: Completed | Type: Observational
Sponsor: Marie-laure Welter (Other)
Responsible Party: Sponsor-Investigator, Marie-laure Welter, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Organization: Groupe Hospitalier Pitie-Salpetriere (Other)
Other Study IDs: P031201
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Basal Ganglia Lesions
Keywords: basal ganglia; loss of psychic self-activation
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Magnetic resonance imaging

SUMMARY:
Basal ganglia are involved in the control of motor, cognitive and emotional behaviours. The aim of this study is to precisely evaluate patients with basal ganglia focal lesions both with or without loss of psychic-self activation.

ELIGIBILITY:
Inclusion Criteria:

* Basal ganglia lesions

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Dementia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lesion of the basal ganglia structures
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2005-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, MD, PhD, Principal Investigator — Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Centre d'Investigation Clinique-Hôpital Pitié-Salpetriere, Paris, France